CLINICAL TRIAL: NCT01315223
Title: Outpatient Lung Impedance-Guided Preventive Therapy in Patients With Chronic Heart Failure (CHF)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0010-11-HYMC
Record Dates: First submitted 2011-03-13; First posted 2011-03-15 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Congestive Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional treatment CHF patients (No Intervention): One hundred and fifty patients with CHF will be treated according to current guidelines (conventional treatment).
- Lung impedence-guided treatment (Experimental)
  Interventions: Other: Lung impedence-guided treatment

INTERVENTIONS:
Other: Lung impedence-guided treatment — One hundred fifty patients with CHF will be treated according to common practice and values of lung impedance
  Arms: Lung impedence-guided treatment

SUMMARY:
Patients suffering from Chronic Heart Failure (CHF) are hospitalized for acute heart failure (AHF) several times a year. Currently, we have no method for prediction of future developments of AHF. In our center we have investigated the monitoring of lung impedence as a predictor for future deterioration. It was found that a decrease in lung impedence of more than 15% from normal value predicts AHF development with sensitivity of 98%. In this study we try to prove the hypothesis that preventive treatment according to lung impedence value may prevent future hospitalizations for AHF and improve clinical outcome.

Patients recruited by year:

2011 - 50; 2012 - 25; 2013 - 35; 2014 - 30; 2015 - 50; 2016 - 5

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from CHF, NYHA II-IV class
* LV lower than 35% to LV lower than 45%

Exclusion Criteria:

* Patients with additional disease with life-expectancy of less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-03; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Reduction of hospitalization for acute heart failure | Five years

SECONDARY OUTCOMES:
Improved clinical outcome for CHF patients | Five years

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Derived] Kleiner Shochat M, Fudim M, Kapustin D, Kazatsker M, Kleiner I, Weinstein JM, Panjrath G, Rozen G, Roguin A, Meisel SR. Early Impedance-Guided Intervention Improves Long-Term Outcome in Patients With Heart Failure. J Am Coll Cardiol. 2021 Oct 26;78(17):1751-1752. doi: 10.1016/j.jacc.2021.08.036. No abstract available. PMID 34674821
- [Derived] Shochat MK, Shotan A, Blondheim DS, Kazatsker M, Dahan I, Asif A, Rozenman Y, Kleiner I, Weinstein JM, Frimerman A, Vasilenko L, Meisel SR. Non-Invasive Lung IMPEDANCE-Guided Preemptive Treatment in Chronic Heart Failure Patients: A Randomized Controlled Trial (IMPEDANCE-HF Trial). J Card Fail. 2016 Sep;22(9):713-22. doi: 10.1016/j.cardfail.2016.03.015. Epub 2016 Apr 4. PMID 27058408